CLINICAL TRIAL: NCT00328419
Title: Consequences of Parenteral Nutrition Photoprotection on the Oxidant Related Diseases Among Extremely Low Birth Weight Infants : A Randomized Controlled Study
Brief Title: Consequences of Parenteral Nutrition Photoprotection on Oxidant Related Diseases Among Extremely Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2004.358
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2011-12

CONDITIONS: Infant, Premature
Keywords: Photoprotection,; Parenteral nutrition; Oxidant stress; Infant, Premature
MeSH Terms: conditions — Premature Birth; Hyperphagia | interventions — Syringes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): photoprotected parenteral nutrition
  Interventions: Device: photoprotected bags, tubing, syringes
- 2 (Active Comparator): Non-photoprotected parenteral nutrition
  Interventions: Device: standard tubing and bags

INTERVENTIONS:
Device: photoprotected bags, tubing, syringes — use of photoprotected parenteral nutrition device
  Arms: 1
Device: standard tubing and bags — Use of standard (transparent) parenteral nutrition device
  Arms: 2

SUMMARY:
The antioxidant system of very low birth weight infants is immature. This immaturity is implicated in the pathogenesis of diseases such as bronchopulmonary dysplasia or retinopathy. The main source of oxidant is oxygen, and parenteral nutrition is contaminated with oxidant. Photoprotection decreases the oxidant load infused with parenteral nutrition. In a preliminary study, photoprotection reduced the frequency of pulmonary bronchodysplasia, increased the quantity of enteral nutrition tolerated, and decreased the arterial blood pressure among very low birth weight infants. The aim of this study is to evaluate the impact of photoprotection on oxidant related diseases among very low birth weight infants. This study is a randomized multicenter trial. In the intervention group, photoprotection is applied until the infusion of parenteral nutrition with amber bags, tubing, and syringes. The quality of photoprotection is controlled by measuring malondialdehyde and cysteine after 24 hours of infusion. The control group will receive parenteral nutrition with transparent bags and tubing. The outcomes are evaluated at 36 weeks, and 680 infants will be enrolled, with stratification among centers and gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 30 weeks gestational age
* Postnatal age between 1 and 6 days
* Apgar score up to 2

Exclusion Criteria:

* Severe congenital abnormalities
* Intraventricular hemorrhage grade up to 2
* Proven sepsis before inclusion
* Transfusion before inclusion
* Use of intravenous lipids or parenteral nutrition before randomisation

Ages: 1 Day to 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 591 (Actual)
Dates: Start 2006-05; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Death or bronchopulmonary dysplasia at 28 days | 28 days

SECONDARY OUTCOMES:
Retinopathy of prematurity | 36 weeks
sepsis | 28 days and 36 weeks
intraventricular hemorrhage | 7 days, 24days, 36 weeks
periventricular leucomalacia | 36 weeks
tolerance of enteral nutrition | during enteral nutrition
enterocolitis | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Laborie, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Angelique Denis, Lyon, France

REFERENCES:
- [Result] Laborie S, Denis A, Dassieu G, Bedu A, Tourneux P, Pinquier D, Kermorvant E, Millet V, Klosowski S, Patural H, Clamadieu C, Brunhes A, Walther M, Jaisson-Hot I, Mandy B, Claris O. Shielding Parenteral Nutrition Solutions From Light: A Randomized Controlled Trial. JPEN J Parenter Enteral Nutr. 2015 Aug;39(6):729-37. doi: 10.1177/0148607114537523. Epub 2014 Jun 12. PMID 24925504